CLINICAL TRIAL: NCT06455410
Title: GP Plus Adebrelimab Versus GP Neoadjuvant Chemotherapy Followed by Concurrent Chemoradiotherapy for High-risk Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: GP Plus Adebrelimab Versus GP Neoadjuvant Chemotherapy for Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, MD, PhD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-FXY-154
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP combined with adebrelimab neoadjuvant therapy+CCRT (Experimental): Adebrelimab (1200mg) to be administered on Day 1 of the Lead-in Phase (-14 days to the start of the neoadjuvant chemoimmunotherapy phase). Patients receive neoadjuvant therapy with gemcitabine (1000mg per square meter on day 1,8) , cisplatin (80mg per square meter on day 1) and adebrelimab (given 1200mg on day 1) every three weeks for three cycles before radiotherapy, then followed by concurrent IMRT and cisplatin (100mg per square meter) concurrent every three weeks during radiotherapy (D1, D22, D43 of RT).
  Interventions: Drug: GP; Drug: Adebrelimab; Drug: concurrent chemoradiotherapy (CCRT)
- GP neoadjuvant therapy+CCRT (Active Comparator): Patients receive neoadjuvant therapy with gemcitabine (1000mg per square meter on day 1,8) , cisplatin (80mg per square meter on day 1) every three weeks for three cycles before radiotherapy, then followed by concurrent IMRT and cisplatin (100mg per square meter) concurrent every three weeks during radiotherapy (D1, D22, D43 of RT).
  Interventions: Drug: GP; Drug: concurrent chemoradiotherapy (CCRT)

INTERVENTIONS:
Drug: GP — gemcitabine + cisplatin
Drug: Adebrelimab — a PD-L1 inhibitor
  Arms: GP combined with adebrelimab neoadjuvant therapy+CCRT
Drug: concurrent chemoradiotherapy (CCRT) — concurrent chemoradiotherapy (CCRT)

SUMMARY:
The purpose of this study is to explore the efficacy and safety of neoadjuvant GP chemotherapy plus adebrelimab versus neoadjuvant GP chemotherapy in treating high-risk locoregionally advanced nasopharyngeal carcinoma patients.

DETAILED DESCRIPTION:
Platinum-based neoadjuvant chemotherapy plus concurrent chemoradiotherapy (CCRT) is the standard of care for patients with locoregionally advanced nasopharyngeal carcinoma (NPC). Gemcitabine plus cisplatin(GP) has been demonstrated an effective chemotherapy regimen for NPC patients in previous studies. Three cycles of GP neoadjuvant chemotherapy resulted in 10% of complete response rate, and GP neoadjuvant chemotherapy added to chemoradiotherapy significantly improved recurrence-free survival (85.3% vs 76.5%) and overall survival (94.6% vs 90.3%) among locoregionally advanced NPC patients , as compared with concurrent chemoradiotherapy alone. Therefore, GP has been established as the highest level of evidence-based neoadjuvant chemotherapy regimen in the 2020 National Comprehensive Cancer Network (NCCN) guidelines. Recently, immune checkpoint inhibitors, such as anti-programmed cell death-1 (PD-1) monoclonal antibody has shown promising efficacy in NPC patients. Clinical trials have shown objective response rates of 20.5%-34% in patients with recurrent or metastatic NPC patients receiving anti PD-1 monoclonal antibody immunotherapy including pembrolizumab, nivolumab, camrelizumab, and toripalimab. GP chemotherapy combined with anti PD-1 antibody were hence considered in treating locoregionally advanced NPC. Concurrent radiotherapy might cause T-cell dysfunction, and larger-volume elective nodal irradiation might hinder immunotherapy effects by directly depleting memory T cells. No survival benefit was observed when PD-1 blockade was added concurrently to the CCRT phase for treating head and neck cancers. On the contrary, several studies have demonstrated that administration of immunotherapy in the neoadjuvant setting modified the primary tumor into an antigen source for T-cell expansion and priming, thereby resulting in stronger effects than those of adjuvant therapy. Currently there were 3 trials exploring the addition of immunotherapy to chemoradiotherapy, the preliminary results of which were recently published. These trials had different trial designs, with two trials utilized anti PD-1 inhibitors in all treatment phases including neoadjuvant, concurrent and adjuvant phases, The third trial, which was conducted by our team, gave anti PD-1 inhibitor only in the neoadjuvant phase, and promising efficacy was observed in our study.

Adebrelimab is a recombinant humanized IgG4 monoclonal antibody with specificity for PD-L1. In a phase III clinical trial of extensive stage small-cell lung cancer, the addition of adebrelimab significantly improved the median overall survival compared with the control group (15.3 vs. 12.8，HR 0.72, P=0.0017). So we hypothesize that GP neoadjuvant chemotherapy combined with adebrelimab could further improve the survival of patients with high-risk locoregionally advanced NPC (diagnosed with T4 or N2-3 disease). Therefore, we designed this phase II multi-center randomized controlled trial to evaluate whether GP neoadjuvant chemotherapy combined with adebrelimab plus cisplatin-based CCRT improve the complete response rate of high-risk locoregionally advanced NPC patients compared with GP neoadjuvant chemotherapy plus CCRT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be informed of the investigational nature of this study and give written informed consent.
2. Age ≥ 18 years and ≤65 years, men or non-pregnant women.
3. Patients with histologically confirmed Nonkeratinizing carcinoma of the nasopharynx (differentiated or undifferentiated type, WHO II or III).
4. Tumor staged as T4N0-1M0 or T1-4N2-3M0 (AJCC 8th).
5. No previous anti-tumor treatment.
6. Eastern Cooperative Oncology Group (ECOG) score 0 or 1.
7. Adequate marrow function: White blood cell count (WBC)≥4.0×109 /L, Hemoglobin ≥ 90g/L, Platelet count ≥100×109/L.
8. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), serum total bilirubin (TBIL) ≤2×upper limit of normal (ULN).
9. Adequate renal function: creatinine clearance rate ≥ 60 ml/min or Creatinine ≤ 1.5× upper limit of normal value.

Exclusion Criteria:

1. Patients with recurrent or metastatic nasopharyngeal carcinoma.
2. Histologically confirmed with keratinizing squamous cell carcinoma of the nasopharynx.
3. Prior therapy with radiation or systemic chemotherapy.
4. Women in the period of pregnancy, lactation, or reproductive without effective contraceptive measures.
5. Seropositivity for human immunodeficiency virus (HIV).
6. Known history of other malignancies (except cured basal cell carcinoma or carcinoma in situ of the cervix).
7. Prior exposure to immune checkpoint inhibitors,including anti-PD-1, anti- PD-L1, anti-CTLA-4 antibodies.
8. Patients with immunodeficiency disease or a history of organ transplantation.
9. Received large doses of glucocorticoids, anticancer monoclonal antibodies, or other immunosuppressants within 4 weeks.
10. Patients with severe dysfunction of heart, liver, lung, kidney or marrow.
11. Patients with severe, uncontrolled disease or infections.
12. Received other research drugs or in other clinical trials at the same time.
13. Refuse or fail to sign the informed consent .
14. Patients with other treatment contraindications.
15. Patients with personality or mental disorders, incapacity or limited capacity for civil conduct.
16. Hepatitis B surface antigen (HBsAg) positive and peripheral blood HBV deoxyribonucleic acid (HBV DNA) ≥1000cps/ml or 200 IU/ml.
17. Patients with positive HCV antibody test will only be enrolled in this study if the PCR test for HCV RNA is negative.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2028-06-18 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | 11weeks
  The proportion of patients who achieve complete response after neoadjuvant chemotherapy or chemoimmunotherapy as assessed by RECIST 1.1.

SECONDARY OUTCOMES:
Event-free survival(EFS) | 2 years
  defined as the time from randomisation to documented locoregional relapse /distant metastasis or death due to any cause, whichever occurred first.
Overall survival (OS) | 2 years
  defined as the time from randomisation to death due to any cause.
Locoregional relapse-free survival（LRRFS） | 2 years
  defined as the time from randomisation to documented locoregional relapse or death due to any cause.
Distant metastasis-free survival (DMFS) | 2 years
  defined as the time from randomisation to documented distant metastasis or death due to any cause
Toxicity profiles | Up to 2 years
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events (acute toxicity) and late radiation toxicities were assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Foshan First People's Hospital, Foshan, Guangdong
  - Affiliated cancer hospital and institute of guangzhou medical university, Guangzhou
  - Sun Yat-Sen Memorial Hospital, Guangzhou
  - The affiliated panyu central hospital of guangzhou medical university, Guangzhou
  - ZhuJiang Hospital of Southern Medical University, Guangzhou
  - Liuzhou Workers Hospital, Liuchow
  - Guangxi Medical University Affiliated Cancer Hospital, Nanning
  - Cancer hospital of Shantou university medical college, Shantou
  - Cancer hospital Chinese academy of medical sciences, Shenzhen center, Shenzhen
  - The second people's hospital of Shenzhen, Shenzhen
  - The university of Hongkong - Shenzhen hospital, Shenzhen
  - Guangdong Medical School First Affiliated Hospital, Zhangjiang